CLINICAL TRIAL: NCT03643133
Title: Multicentre, Randomised, Phase 2 Trial of Mifamurtide Combined With Post-operative Chemotherapy for Newly Diagnosed High Risk Osteosarcoma Patients (Metastatic Osteosarcoma at Diagnosis or Localised Disease With Poor Histological Response)
Brief Title: Mifamurtide Combined With Post-operative Chemotherapy for Newly Diagnosed High Risk Osteosarcoma Patients
Acronym: SARCOME13
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-0150/1704; 2017-001165-24 (EudraCT Number)
Record Dates: First submitted 2018-07-11; First posted 2018-08-22 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Osteosarcoma
Keywords: Bone; Neoplasm, bone tissue; Acetylmuramyl-Alanyl-Isoglutamine
MeSH Terms: conditions — Osteosarcoma; Neoplasms, Bone Tissue | interventions — mifamurtide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Active Comparator): Post-operative chemotherapy alone (EI or M-API regimen depending on patient age) :
  M-API regimen (≤25 years) :
  Doxorubicin 60 mg/m², Day 1 Ifosfamide 3 g/m² Day 1 and 2 Cisplatin 100 mg/m², Day 2
  EI regimen (26-50 years) :
  Etoposide 75 mg/m²/d, Day 1-4 Ifosfamide 3 g/m²/d, Day 1-4
  Interventions: Combination Product: EI or M-API regimen depending on patient age
- Experimental arm (Experimental): Post-operative chemotherapy (EI or M-API regimen) combined with Mifamurtide 2 mg/m² twice weekly post-randomisation for 12 weeks then weekly for 24 weeks
  Interventions: Drug: Mifamurtide; Combination Product: EI or M-API regimen depending on patient age

INTERVENTIONS:
Drug: Mifamurtide — 48 doses overall over 36 weeks
  Other Names: MEPACT
  Arms: Experimental arm
Combination Product: EI or M-API regimen depending on patient age — M-API regimen:
  One course of high-dose Methotrexate (optional) followed by 5 courses of API, every 21 days
  EI regimen :
  5 course of EI, every 21 days

SUMMARY:
Trial evaluating the impact on efficacy of mifamurtide as add-on treatment to post-operative chemotherapy compared to post-operative chemotherapy alone in first-line treatment of patients with high-risk osteosarcoma (defined as metastatic osteosarcoma at diagnosis or localised osteosarcoma with poor histological response).

DETAILED DESCRIPTION:
Multicentre, randomised, open-label, phase II trial, with 2 parallel groups. After pre-operative chemotherapy and surgery of the primary tumour and lung metastases (if applicable), patients presenting high-risk osteosarcoma (defined as metastatic osteosarcoma at diagnosis or localised osteosarcoma with poor histological response) will be randomised between 2 arms:

* Control arm: post-operative chemotherapy alone (with regimens adapted to the age of patient)
* Experimental arm : post-operative chemotherapy combined with mifamurtide

This randomised trial is part of a study recruiting all patients ≤50 years old with a newly diagnosed high-grade osteosarcoma.

ELIGIBILITY:
Registration Criteria:

1. All newly diagnosed, biopsy-proven, high-grade osteosarcoma, whatever the initial extension of the disease
2. Age >2 years and ≤50 years;
3. Normal haematological, renal, cardiac and hepatic functions
4. Planned neoadjuvant chemotherapy as follows:

   1. Methotrexate-Etoposide-Ifosfamide (M-EI regimen) for patients ≤25 years
   2. Doxorubicin-Cisplatin-Ifosfamide (API-AI regimen) for patients 26-50 years
5. Written informed consent from patients and/or their parents/guardians before enrolment and any study-related procedure
6. Affiliation to a social insurance regimen

Inclusion Criteria:

1. Patient with a histologically proven, confirmed by experts pathologists panel (before surgery at the latest), high-grade osteosarcoma
2. Registered at diagnosis into the study
3. Primary tumour resected after pre-operative chemotherapy
4. Osteosarcoma classified as high risk because of at least one risk factor:

   1. presence of distant metastases or skip metastases at diagnosis
   2. and/or poor histological response to pre-operative chemotherapy (>10% residual viable cells on the analysis of the primary tumour surgical specimen)
5. Pre-operative chemotherapy combining

   1. Methotrexate-Etoposide-Ifosfamide (M-EI regimen) for patients ≤25 years
   2. Doxorubicin-Cisplatin-Ifosfamide (API-AI regimen) for patients 26-50 years
6. Screening laboratory values must meet the following criteria (using CTCAE v4) and should be obtained within 7 days prior to randomisation:

   1. Absolute neutrophil count ≥1.0 x 10⁹/L
   2. Platelets ≥100 x 10⁹/L
   3. Haemoglobin ≥8.0 g/mL
   4. Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤2.5 x upper limit of normal (ULN) in the absence of liver metastases or ≤5 x ULN in the presence of liver metastases
   5. Total Bilirubin ≤2 x ULN (except Gilbert Syndrome: <3.0 mg/dL) or Total Bilirubin ≤5.0 x ULN in the presence of liver metastases
   6. Creatinine clearance ≥60 mL/min/1.73 m² according to the Schwartz or Cockcroft formula according to patient's age
7. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) done within 7 days prior to randomisation
8. Provision of dated and signed written informed consent for the randomised trial prior to any study specific procedures, sampling and analyses.
9. Patient fit to undergo protocol treatment and follow-up
10. Affiliation to a social insurance regimen

Exclusion Criteria:

1. Low grade osteosarcoma, parosteal or periosteal osteosarcoma
2. Prior history of other malignancies other than study disease (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix) unless the patient has been free of the disease for at least 3 years.
3. Osteosarcoma with multiple metastases for whom complete removal is not expected to be feasible even after shrinkage with chemotherapy
4. Progressive disease at any site under initial chemotherapy, confirmed before randomisation time, and not totally resected during surgery
5. Any medical condition precluding treatment with protocol chemotherapy
6. Fractional Shortening <28% or left ventricular ejection fraction (LVEF) 50% before treatment (only for API post-operative chemotherapy) by echocardiogram or multigated acquisition (MUGA) scan
7. Pregnancy or breast-feeding
8. Hypersensitivity to the active substance or to any of the excipients
9. Concurrent use of immunodepressive treatment such as cyclosporine, tacrolimus or other calcineurin inhibitors
10. Concurrent use with high-dose non-steroidal anti-inflammatory drugs (NSAIDs, cyclooxygenase inhibitors)
11. Inflammatory or auto-immune disease, allergy or asthma requiring a chronic use of steroid treatment that cannot be stopped.
12. Patients with positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
13. Patients with positive tests for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating active or chronic infection.

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2033-10 (Estimated)

PRIMARY OUTCOMES:
Compare event-free survival in the treatment arms | Expected average duration of 3 years from randomization
  Event-free survival defined as the time duration from randomisation to time of first event (loco-regional or distant relapse or progression, second malignancy, death from any cause)

SECONDARY OUTCOMES:
Compare overall survival in the treatment arms | Up to 10 years from randomization
  Overall survival defined as the time duration from randomisation to death, whatever the cause of death
Compare actual and planned cumulative dose and dose intensity of mifamurtide | Up to 36 weeks from randomization (until end of treatment)
  Calculation of actual cumulative dose and dose intensity compared to the planned treatment administration schedule
Compare the incidence of adverse events in the treatment arms | Up to 40 weeks from randomization (4 weeks after end of treatment)
  Evaluation of toxicity (graded by NCI-CTCAE v4)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie MD GASPAR, PhD, Principal Investigator — Gustave Roussy Cancer Campus; Sophie MD PIPERNO-NEUMANN, PhD, Principal Investigator — Institut Curie
Locations (31):
- France (31):
  - CHU Amiens-Picardie - Service d'oncologie hématologie pédiatrique, Amiens
  - CHU d'Angers - Service d'oncologie pédiatrique, Angers
  - Institut Bergonié - Service d'oncologie médicale, Bordeaux
  - CHU de Caen - Service d'oncologie hématologie pédiatrique, Caen
  - CHU de Grenoble - Service d'oncologie hématologie pédiatrique, La Tronche
  - Centre Oscar Lambret - Unité d'onco-pédiatrie, Lille
  - Centre Léon Bérard - IHOPE, Lyon
  - Centre Léon Bérard - Service d'oncologie médicale, Lyon
  - Hôpital de la Timone - service d'oncologie médicale, Marseille
  - Hôpital de la Timone - Service d'oncologie pédiatrique, Marseille
  - CHU Arnaud de Villeneuve - Onco-hématologie pédiatrique, Montpellier
  - Institut régional du Cancer de Montpellier - Service d'oncologie médicale, Montpellier
  - CHU de Nantes - Service d'oncologie hématologie pédiatrique, Nantes
  - CHU de Nice - Service d'oncologie hématologie pédiatrique, Nice
  - Institut Curie - Service d'oncologie médicale, Paris
  - Hôpital Armand Trousseau - Service d'hématologie et d'oncologie pédiatrique, Paris
  - Hôpital Cochin, Paris
  - Institut Curie - Service d'oncologie pédiatrique, Paris
  - Centre Eugène Marquis - Service d'oncologie médicale, Rennes
  - Hôpital Charles Nicolle - Hémato-Immuno-Oncologie Pédiatrique, Rouen
  - Institut de Cancérologie de l'Ouest (Site René Gauducheau) - Service d'oncologie médicale, Saint-Herblain
  - Hôpital de Hautepierre - Onco-hématologie adulte, Strasbourg
  - Hôpital Hautepierre - Onco-hématologie pédiatrique, Strasbourg
  - CHU Toulouse - Hôpital des Enfants - Service d'Hémato-Immuno-Oncologie, Toulouse
  - Institut Claudius Regaud - service d'oncologie médicale, Toulouse
  - CHU Bretonneau - Service d'oncologie médicale, Tours
  - Hôpital Clocheville - Hématologie et oncologie pédiatrique, Tours
  - CHRU de Nancy - Onco-hématologie pédiatrique, Vandœuvre-lès-Nancy
  - Institut de Cancérologie de Lorraine - Service d'oncologie médicale, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy - Service de cancérologie de l'enfant et de l'adolescent, Villejuif
  - Institut Gustave Roussy - Service d'oncologie médicale, Villejuif

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared at an individual level, they will be part of the study database including all enrolled patients.

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903
- [Derived] Brard C, Piperno-Neumann S, Delaye J, Brugieres L, Hampson LV, Le Teuff G, Le Deley MC, Gaspar N. Sarcome-13/OS2016 trial protocol: a multicentre, randomised, open-label, phase II trial of mifamurtide combined with postoperative chemotherapy for patients with newly diagnosed high-risk osteosarcoma. BMJ Open. 2019 May 19;9(5):e025877. doi: 10.1136/bmjopen-2018-025877. PMID 31110092